CLINICAL TRIAL: NCT00598260
Title: Active Management Of Risk In Pregnancy At Term - a Prospective Study
Brief Title: Active Management Of Risk In Pregnancy At Term to Reduce Rate of Cesarean Deliveries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Shai Pri-Paz, Albert Einstein Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: (H)N-2957
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Pregnancy
Keywords: active management; induction of labor; cesarean delivery; Cesarean
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- study group (Experimental): study group - induction of labor at optimal time of delivery between 38 weeks and 41 weeks.
  Interventions: Procedure: induction of labor
- 2 - control group (No Intervention): control group

INTERVENTIONS:
Procedure: induction of labor — study group - induction of labor at optimal time of delivery between 38 weeks and 41 weeks.
  Arms: 1- study group

SUMMARY:
This is a prospective randomized cohort study of obstetric patients from Paley clinic at AEMC and from other affiliated obstetric clinics.

This study will try to determine if active management of risks in pregnancy at term by inducing patients will not decrease the cesarean delivery rate or change neonatal outcomes.

The outcomes that will be measured include cesarean delivery rate, meconium, Apgar scores and admissions to the NICU.

DETAILED DESCRIPTION:
The study will include patients who have their prenatal care at the Paley clinic in AEMC, where the residents provide the prenatal care with supervision of OBGYN attending physicians, or at other affiliated clinics that are staffed by care givers from our OBGYN department.

Patients at our obstetric clinics are scheduled for weekly visits starting at 36 weeks. At 36 to 37 weeks of gestation, or earlier, each patient will be offered to participate in the study. Those who refuse will continue to have the standard care and will not be considered as part of the study. Those who wish to participate in the study will be consented and will then be randomly assigned to the control group or to the AMOR-IPAT group with a ratio of 2:1.

Risk factors will be identified for each patient participating in the study at the gestational age of 36 to 37 weeks (using the digichart system, the medical records and questioners) and the upper limit of the optimal time of delivery will be calculated for each patient, according to the method used by the UPenn group, with the time always being at least 38 weeks and no more then 41 weeks.

Patients from the AMOR-IPAT group will be scheduled for induction of labor on the morning of the day of the calculated upper limit (plus or minus 2 days).

To try and eliminate biases, a uniform method of induction will be applied to all the patients participating in the study, no matter the group or the reason for the induction. The induction will be performed with misoprostol 25mcg intravaginally every four hours (to a maximum of three doses) for a Bishop score of 4 or less and as long as there is no tachysystole which will be defined as six or more uterine contractions in ten minutes in consecutive ten minute intervals. The misoprostol will be followed by a foley bulb inflated with 80 cc of fluid if the cervix is still not favorable after three doses or when tachysystole develops. Once the cervix is favorable induction will be continued with high dose oxytocin (starting dose of six milliunits with increments of four milliunits every thirty minutes), which is associated with less cesarean deliveries for dystocia than the low dose.

Anesthesia will be applied according to the patient's wish, without limiting epidural anesthesia to a certain degree of dilatation.

After delivery information will be collected from the charts and the two groups will be compared regarding the incidence of cesarean deliveries, but also regarding intrapartum variables and major outcomes.

The Student t test and the Wilcoxon rank sum test will be used to compare continuous demographic characteristics, past medical and surgical historic features and obstetric risk factors that will be present in the two study groups. Universal chi squared tests will be used to compare levels of various dichotomous variables.

Statistical significance is defined as a probability value of less than 0.05. Using a power analysis and by assuming a cesarean delivery rate of 20% in the control group and a change of 13% (as shown in the original study) we will need 191 patients in the control group and 96 in the study group.

All data will be collected by staff of the OBGYN department and maintained on departmental secured password limited database. Obstetrical prenatal data is maintained on HIPPA compliant password protected electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* patients with singleton pregnancies
* at least one prenatal visit at one of our clinics
* an ultrasonogram confirming the dates within the first 22 weeks
* no maternal or fetal problems before 37 weeks and 5 days of gestation that mandated cesarean delivery.

Exclusion Criteria:

* a delivery before 37 weeks and 5 days of gestation
* a previous cesarean delivery (one or more)
* a history of any other uterine surgeries that are a contraindication for a vaginal delivery.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 222 (Actual)
Dates: Start 2006-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
cesarean delivery rate | prospective: 06.2006 to 06.2008

SECONDARY OUTCOMES:
admissions to NICU during same hospitalization | prospective. 06.2006 - 06.2008
APGAR scores at one and five minutes | prospective. 06.2006 - 06.2008
meconium | prospective. 06.2006 - 06.2008

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Cohen, MD, Study Chair — Albert Einstein Medical Center; Shai M Pri-Paz, MD, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States